CLINICAL TRIAL: NCT04514705
Title: Clinical Respiratory Investigation in Post Covid-19 Patients
Brief Title: Characteristics in Post Covid-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Director of Human Movement Department, Universidade Metodista de Piracicaba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F110820
Record Dates: First submitted 2020-08-11; First posted 2020-08-17 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Coronavirus Infection
Keywords: Rehabilitation; Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Exercise
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): The exercises performed will attend the musculoskeletal dimension of the body, which includes the muscular strength / endurance indexes, which is part of the functional-motor dimension of physical fitness related to health. The protocol will be applied in the form of sessions lasting approximately 50 minutes, performed three times a week on alternate days, for a period of 6 weeks, totaling 20 sessions. For aerobic exercises, a treadmill will be used and for anaerobic exercises, four exercises involving muscle mobility / strength in upper and lower limbs will be performed at weight training station.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise with treadmil and weight training station

SUMMARY:
To evaluate pulmonary changes and the results of a cardiopulmonary rehabilitation protocol (CPRP) in patients after SARS-VOC-2 infection. Clinical trial type study to be conducted between 2020 and 2024 involving clinical-functional cardiopulmonary imaging and blood transcriptome profile: before CPRP (T1), 2 months after CPRP (T2) and 1 year later (T3). Expected results: a) clinical, image and transcriptome changes; b) clinical-functional improvement after CPRP.

ELIGIBILITY:
Inclusion Criteria:

* With confirmed diagnosis for SARS-COV-2.

Exclusion Criteria:

* With any type of simultaneous pneumopathy.
* Patients with autoimmune disease
* People with simultaneous infectious diseases
* Pregnant women
* With degenerative diseases of the nervous system or musculoskeletal system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Characteristics of lung | post treatment in 3 days
  In the supine position, the patient will perform deep inspiration followed by momentary apnea inside the high resolution scanner to capture cross-sectional images of the chest with smaller cuts than 1mm of collimation which helped in the detection of even small lesions.
Respiratory muscle strength | post treatment in 3 days
  Respiratory muscle strength will be assessed using the digital manovacuometer. The measurement will be performed as follows the patient will be asked to empty the lungs to the residual volume and then perform an inhalation until the total lung capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade do Estado do Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kamalakannan S, Chakraborty S. Occupational therapy: The key to unlocking locked-up occupations during the COVID-19 pandemic. Wellcome Open Res. 2020 Jul 1;5:153. doi: 10.12688/wellcomeopenres.16089.1. eCollection 2020. PMID 32766458
- [Result] Torlinski T, Rakasz L, Wysota B, Czyz M, Snelson C. An interdisciplinary approach to the management of critically ill patients during covid-19 pandemic; an experience of a university hospital in England. Wiad Lek. 2020;73(7):1576-1579. PMID 32759457
- [Result] Rooney S, Webster A, Paul L. Systematic Review of Changes and Recovery in Physical Function and Fitness After Severe Acute Respiratory Syndrome-Related Coronavirus Infection: Implications for COVID-19 Rehabilitation. Phys Ther. 2020 Sep 28;100(10):1717-1729. doi: 10.1093/ptj/pzaa129. PMID 32737507
- [Result] Saeki T, Ogawa F, Chiba R, Nonogaki M, Uesugi J, Takeuchi I, Nakamura T. Rehabilitation Therapy for a COVID-19 Patient Who Received Mechanical Ventilation in Japan. Am J Phys Med Rehabil. 2020 Oct;99(10):873-875. doi: 10.1097/PHM.0000000000001545. PMID 32732744
- [Result] Grigoletto I, Cavalheri V, Lima FF, Ramos EMC. Recovery after COVID-19: The potential role of pulmonary rehabilitation. Braz J Phys Ther. 2020 Nov-Dec;24(6):463-464. doi: 10.1016/j.bjpt.2020.07.002. Epub 2020 Jul 19. No abstract available. PMID 32723665
- [Result] Abdullahi A, Bello B, Mukhtar NB, Kaka B, Abba MA, Usman JS, Shittu A, Mayana KI, Maiwada SA, Mohammed J. Physiotherapy management of COVID-19 in Africa: Ongoing efforts, challenges, and future directions. Physiother Theory Pract. 2020 Aug;36(8):871-872. doi: 10.1080/09593985.2020.1798163. Epub 2020 Jul 29. No abstract available. PMID 32723204